CLINICAL TRIAL: NCT01346566
Title: Cionni Ring and In-the-bag IOL Implantation for Subluxated Lenses: A Prospective Case Series
Brief Title: Prospective Study of Cionni Ring and In-the-bag IOL Implantation for Subluxated Lenses
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Iladevi Cataract and IOL Research Center (Other)
Responsible Party: Dr. Abhay R. Vasavada, Iladevi Cataract and IOL Research Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICIRCcionni
Record Dates: First submitted 2011-04-30; First posted 2011-05-03 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Lens Subluxation
Keywords: Cionni Ring; In-the-bag IOL; Subluxated lenses; Intraoperative Performance; Postoperative Outcome
MeSH Terms: conditions — Lens Subluxation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Cionni Modified Capsule Tension Ring — Cionni ring was used to fixate the capsular bag to the sclera and IOL was implanted in-the-bag

SUMMARY:
The purpose of this study is to report the intraoperative performance and postoperative outcomes of the Cionni-modified capsule tension ring implantation in eyes with subluxated lenses.

DETAILED DESCRIPTION:
The introduction of endocapsular stabilising devices have significantly improved the management of zonular weakness, allowing for in-the-bag IOL implantation. The Cionni modified capsule tension ring (M-CTR) has an anterior eyelet that provides for fixation of the capsular bag without violating its integrity. Adult and pediatric studies have shown the usefulness of the M-CTR to manage zonular weakness. However, there are very few prospective studies that show the outcomes following implantation of the M-CTR and in-the-bag IOL on a longterm basis. Therefore, the investigators decided to carry out this study to report the intraoperative performance and postoperative outcomes on a longterm basis following M-CTR and in-the-bag intraocular lens (IOL) implantation.

ELIGIBILITY:
Inclusion Criteria:

* Subluxated Lenses
* Traumatic or Non-traumatic etiology

Exclusion Criteria:

* Dislocated Lenses

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2003-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
IOL Centration | 4 years follow-up

SECONDARY OUTCOMES:
Complications | 4 years follow-up
IOP | 4 years
Posterior Capsule Opacification | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Abhay R Vasavada, MS, FRCS, Principal Investigator — Iladevi Cataract & IOL Research Centre
Locations (1):
- Iladevi Cataract & IOL Research Centre, Ahmedabad, Gujarat, India

REFERENCES:
- [Derived] Vasavada AR, Praveen MR, Vasavada VA, Yeh RY, Srivastava S, Koul A, Trivedi RH. Cionni ring and in-the-bag intraocular lens implantation for subluxated lenses: a prospective case series. Am J Ophthalmol. 2012 Jun;153(6):1144-53.e1. doi: 10.1016/j.ajo.2011.11.012. Epub 2012 Feb 7. PMID 22317913